CLINICAL TRIAL: NCT03632304
Title: The Quality of Recovery of Local Anesthesia With Minimal Sedation and Brachial Plexus Block in Hand Surgery: A Randomized Controlled Study
Brief Title: Local Anesthesia With Minimal Sedation and Brachial Plexus Block in Hand Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Fanyi Meng, Resident, Division of Plastic and Reconstructive Surgery, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018-3814
Record Dates: First submitted 2018-08-08; First posted 2018-08-15 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Hand Surgery; Quality of Recovery; Hand Injuries; Hand Fracture; Hand Tendon Injury; Anesthesia, Local
Keywords: hand surgery; quality of recovery; local anesthesia; regional anesthesia; QoR-15
MeSH Terms: conditions — Hand Injuries | interventions — Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brachial plexus block (infraclavicular) (No Intervention): The standard of care at our institution. Performed by experienced regional anesthetists.
- Local anesthesia with minimal sedation (Active Comparator): The comparison group. Performed by the operating surgeon.
  Interventions: Procedure: Local anesthesia with minimal sedation

INTERVENTIONS:
Procedure: Local anesthesia with minimal sedation — The operating surgeon will perform a digital or wrist block to numb the surgical area prior to the surgery, instead of using a brachial plexus block.
  Arms: Local anesthesia with minimal sedation

SUMMARY:
A major innovation in hand surgery in the last decade is the popularization of Wide Awake Hand Surgery (WAHS). This technique consists of numbing the surgical area with local anesthesia with epinephrine and allowing the patient to actively move their hand intra-operatively to assess the strength and quality of repairs or fixations. Despite its theoretical advantages, the application in clinical practice has seldom spread further than simple hand operations, such as carpal tunnel and trigger finger releases. In many institutions, the current standard of care for hand surgery is the brachial plexus block. The primary objective of the study to directly compare the effects of local anesthesia with minimal sedation, performed by the surgeon, and the brachial plexus block, performed by the anesthesiologist, on patient-reported quality of recovery.

Currently, there are no studies in the surgical literature directly comparing patient-reported quality of recovery, post-operative pain control, or time efficiency between local anesthesia and the brachial plexus block in hand surgery. This lack of information is a major impediment to the acceptance and adoption of a simple yet effective anesthesia technique that may increase patient satisfaction and time efficiency in the operating room. This proposed prospective randomized controlled study will quantitatively compare local anesthesia and brachial plexus block on three fronts: 1) patient-reported recovery at 24-hours post-surgery using the validated Quality of Recovery 15 score (QoR-15), 2) post-operative pain and opioid use at 24-hours post-surgery, and 3) nonsurgical time (defined as the time elapsed from one surgery's end time to the next surgery's start time) as a metric for turnover efficiency. The investigators hypothesize that patients randomized to the local anesthesia group will have a more positive recovery experience, a similar pain profile compared to the brachial plexus block despite common beliefs, and a shorter anesthesia-related and nonsurgical time.

The importance of patient-centered care cannot be understated in a successful and high-quality health care system. The results of this study will provide valuable information regarding the patient experience during their post- operative recovery.

DETAILED DESCRIPTION:
In many hospitals, the widely-accepted benefits of local anesthesia have moved minor hand operations such as carpal tunnel and trigger finger release outside of the main operating room. The proven benefits of local anesthesia include increased efficiency, convenience and patient comfort, reduced costs, lack of pre-operative tests, and decreased operative time. Multiple complex hand operations have been described using lidocaine and epinephrine only, with the patient wide awake during surgery. These include K-wire fixation, flexor tendon repair, tendon transfers, and tendon grafting. For those unfamiliar with this technique, the main concerns are that it is poorly tolerated, does not prevent patient movement, and inadequately controls post-operative pain, which all negatively influence a surgeon's comfort and adoption of this technique. Thus, despite its many advantages, local anesthesia in complex hand surgery is still not widely practiced in North America.

Alternatively, the brachial plexus block is a common method of regional anesthesia used in hand surgery, consisting of anesthetizing the entire upper limb via local anesthesia infiltration of the brachial plexus. This reliable sensorimotor blockade is performed under ultrasound guidance by an anesthesiologist approximately 30 minutes prior to surgery. Although safe and effective to use, its long duration of action, increased need for operating room resources, and unpleasant sensation of a flaccid and insensate upper extremity has prompted research into alternative ultrasound-guided nerve blocks in hand surgery.

Despite prior published data on the use of local anesthesia with epinephrine and brachial plexus blocks in hand surgery, there is a paucity of randomized-controlled, prospective, patient-reported outcome studies comparing these two methods of anesthesia. This study aims to capture patient-reported quality of recovery using a validated, psychometrically tested questionnaire, the Quality-of-Recovery 15. A recent systematic review of the measurement properties of QoR-15 showed good content validity and internal consistency, and concluded that it fulfills requirements for outcome measurement instruments in clinical trials.

Preliminary data was obtained from a pilot study of 11 hand surgery patients who underwent a brachial plexus block and were called 24 hours after surgery to answer the QoR-15 questionnaire. The computed mean QoR score was 118/150 +/- 15, consistent with values reported in the literature. This pilot study allowed for the calculation of a projected sample size for this study, outlined below.

This is a prospective single institution randomized controlled study taking place at the Montreal General Hospital, in Montreal, Canada. The institution is a level I trauma center which performs a minimum of 250 upper extremity surgeries yearly. The study participants are trauma or elective hand surgery patients above 18 years undergoing surgery less than 2 hours in duration distal to the carpal bones.

Patients who consent to the study will be randomized to receive local anesthesia with minimal sedation (intervention group) or a brachial plexus block (control group) using www.random.org, a random number generating website. The local anesthesia in the intervention group will be administered by the operating hand surgeon or a senior resident under the surgeon's direct supervision as a wrist block and/or digital block. The regional blocks in the control group will be performed as an infraclavicular brachial plexus block by a staff anesthesiologist with extensive experience in ultrasound-guided regional anesthesia.

This study is designed as a prospective non-inferiority study using an alpha of 0.05 for statistical significance and a power of 80%. Using QoR-15 values derived from the pilot study with effect size of 0.54, a power analysis was conducted, yielding a sample size of 44 patients per group, for a total of 88 patients. All quantitative outcome parameters will be evaluated for normal distribution and reported as mean +/- SD or median (IQR). Differences between two groups will be evaluated using unpaired Student's T-Test (if parametric) or Mann-Whitney-U test (if non-parametric).

The patients will be called on the first post-operative day, at least 24 hours after the end of their surgery, by a research assistant blinded to the randomization. As a primary outcome measure, the patient will be asked to answer the questions on the QoR-15 without revealing their surgery or method of anesthesia. The dosage of the medications used and the number of times an opioid medication was taken will be recorded. The nonsurgical time for the local anesthesia and brachial plexus groups will also be directly compared. Nonsurgical time is defined as the time elapsed between the completion of surgical closure on one case until the surgical incision on the next case.

The study will be conducted in accord with the Tri-Council Policy Statement: Ethical Conduct for Research Involving Humans (2014) as well as in respect of the requirements set out by the McGill University Health Centre Research Ethics Board.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 and older
* Hand surgeries distal to carpal bones
* Trauma and elective cases
* Under 2 hours estimated surgical duration
* Consents to research

Exclusion Criteria:

* Patient refusal
* Allergy to local anesthetics
* Surgery proximal to the carpal bones
* BMI > 40 kg/m2
* Non-compressive neurological disease of the upper extremity
* Daily use of opioids for greater than 2 weeks prior to surgery
* History of complex regional pain syndrome (CRPS)
* Patients with high anxiety or severe post-traumatic stress disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery 15 Questionnaire (QoR-15) | At 24 hours post-surgery
  This psychometrically tested and validated 15-items questionnaire measures patient-reported quality of recovery from surgery and anesthesia on the first post-operative day. Each item consists of a question related to the patient's post-operative recovery and is rated by the patient on a 10-point scale, where 0 means "none of the time" and 10 means "all of the time". The total combined score is obtained from the summation of 15 sub-scores and ranges from 0 to 150, and is used to assess and compare the patient's quality of recovery quantitatively between different interventions. A higher number on the score indicates an improved patient recovery experience. This scale has been validated in the ambulatory surgery setting.

SECONDARY OUTCOMES:
Block performance time, onset time, and nonsurgical time | Within 24 hours of surgery
  To compare local anesthesia to brachial plexus block in hand surgery with respect to performance time, onset time, and nonsurgical time.
Opioid use at 24 hours after surgery | At 24 hours post-surgery
  To evaluate patient-reported 24-hours post-operative pain and use of opioid analgesia following local anesthesia versus brachial plexus block.

CONTACTS AND LOCATIONS:
Overall Officials: Fanyi Meng, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (2):
- Canada (2):
  - Montreal General Hospital, Montreal, Quebec
  - St-Mary's Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No
There will be no need to share individual participant data based on the objectives set out by our research.

REFERENCES:
- [Background] Lalonde DH. Reconstruction of the hand with wide awake surgery. Clin Plast Surg. 2011 Oct;38(4):761-9. doi: 10.1016/j.cps.2011.07.005. PMID 22032599
- [Background] Lalonde D. Minimally invasive anesthesia in wide awake hand surgery. Hand Clin. 2014 Feb;30(1):1-6. doi: 10.1016/j.hcl.2013.08.015. Epub 2013 Nov 9. PMID 24286736
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Background] Soberon JR Jr, Crookshank JW 3rd, Nossaman BD, Elliott CE, Sisco-Wise LE, Duncan SF. Distal Peripheral Nerve Blocks in the Forearm as an Alternative to Proximal Brachial Plexus Blockade in Patients Undergoing Hand Surgery: A Prospective and Randomized Pilot Study. J Hand Surg Am. 2016 Oct;41(10):969-977. doi: 10.1016/j.jhsa.2016.07.092. Epub 2016 Aug 11. PMID 27524691
- [Derived] Meng F, Baradaran A, Jaberi MM, Tran QH, Finlayson R, Luc M, Xu L, Thibaudeau S. Patient-Reported Quality of Recovery after Local Anesthesia versus Brachial Plexus Block in Hand Surgery: A Randomized Controlled Study. Plast Reconstr Surg. 2023 Dec 1;152(6):1287-1296. doi: 10.1097/PRS.0000000000010688. Epub 2023 May 16. PMID 37189224